CLINICAL TRIAL: NCT01530048
Title: A Randomised, Single Centre, Double-blind, Two-period, Cross-over Trial, Assessing the Bioequivalence Between Insulin Aspart 100 U/mL and Insulin Aspart 200 U/mL in Healthy Individuals
Brief Title: Bioequivalence of Two Insulin Aspart Formulations (100 U/mL Versus 200 U/mL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDS290-1750; 2005-005538-11 (EudraCT Number)
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- U200 (Experimental)
  Interventions: Drug: insulin aspart
- U100 (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — A single bolus injection of 0.2 U/kg administered subcutaneously (s.c., under the skin) on two separate dosing visits with a wash-out period 2-15 days in-between

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to test if there is bioequivalence between the insulin aspart 100 U/mL (U100) formulation and the new insulin aspart 200 U/mL (U200) formulation.

ELIGIBILITY:
Inclusion Criteria:

* Considered to be healthy as judged from vital signs, medical history, ECG (electrocardiogram), laboratory values, and physical examination
* Body mass index between 18 and 27 kg/m^2 (both inclusive)
* Non-smoker
* Fasting blood glucose maximum 6 mmol/L
* HbA1c below 6.4%

Exclusion Criteria:

* Pregnant or breast-feeding women
* Women not using acceptable methods of contraception without difficulties for at least three months prior to trial start (screening), including intrauterine devices, oral contraceptives, hormonal implants, or sterilisation
* Clinically significant abnormal laboratory values (as judged by the Investigator)
* Close relative with type 1 diabetes mellitus (father, mother, sister or brother)
* Intake of alcohol within the last 24 hours prior to screening and drug administration visits
* Blood donation or blood loss of more than 500 mL within the 3 last months before screening
* Strenuous exercise within 48 hours before screening as well as drug administration and followup
* Smoking during the past month before drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) in the interval of 0-6 hours
Cmax, maximum concentration

SECONDARY OUTCOMES:
AUC in the interval of 0-infinity hours
tmax, time to reach Cmax
Terminal rate constant
Vz/f, volume of distribution during terminal phase
t½, terminal half-life
AUCGIR, area under the glucose infusion rate value curve
GIRmax, maximum glucose infusion rate value
tGIRmax, time to maximum glucose infusion rate value
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hvidovre, Denmark

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com